CLINICAL TRIAL: NCT06555679
Title: Evaluation of a Predictive Score for the Onset of Moderate to Severe Alcohol Withdrawal Syndrome, the PAWSS, in a Population of Intensive Care Patients at Brest University Hospital
Acronym: PAWSS-ICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0126 PAWSS-ICU
Record Dates: First submitted 2024-08-08; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: prediction; intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
alcohol use disorder (AUD) is a very common condition in patients admitting in ICU's. Brutal stop of alcohol consumption may lead to a withdrawal syndrome, wich is associated with a worse outcome for ICU patients (longuer ICU and hospital stays, use of mechanical ventilation, traumas). The aim of this study is to valid a score (PAWSS : prediction of alcohol withdrawal syndrome (AWS) scale) to predict at admission mild to severe AWS in ICU patients population.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* able to answer to PAWSS in the first 48hours of ICU stay

Exclusion Criteria:

* No alcohol consumption in the last 30 days
* hospital stay of more than 5 days at ICU admission
* hospital stay less than 5 days in total
* expected sedation time of more than 48h
* patient not able to understand the PAWSS
* no consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of PAWSS statistic performances to predict AWS in ICU patients | the first 5 days of hospital stay
  Evaluation of sensitivity, specificity, positive and negative predictive values of PAWSS to predict moderate or severe AWS (defined by a CIWA greater than or equal to 8)

SECONDARY OUTCOMES:
Creation of a new score, the PAWSS-ICU, able to predict AWS in ICU patients | during ICU stay
  To this end, the characteristics of the [no weaning/minimal weaning] and [moderate weaning/severe weaning] groups will be compared, in order to identify significant differences between these two groups, and thus enable the creation of a new score.
  On an exploratory basis :
  * assess the incidence of alcohol misuse and withdrawal syndrome in our population,
  * assess the incidence of complications in the population with moderate to severe withdrawal (trauma, occurrence of pneumopathy, need for mechanical ventilation),
  * assess length of hospital stay and in-hospital mortality.
  Translated with DeepL.com (free version)

OTHER OUTCOMES:
Evaluation of alcohol use disorders (AUD) ans AWS in our population | during ICU stay
  AUD definition for our study :
  * AUD is mentionned in patient's medical record
  * heavy alcohol use (more than 3 drinks a day for a men ant more than 2 drinks a day for a woman)
  * harmful use : physical or psychological complications of alcohol use (liver cirrhosis, depression, ...)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

REFERENCES:
- [Background] Wood E, Albarqouni L, Tkachuk S, Green CJ, Ahamad K, Nolan S, McLean M, Klimas J. Will This Hospitalized Patient Develop Severe Alcohol Withdrawal Syndrome?: The Rational Clinical Examination Systematic Review. JAMA. 2018 Aug 28;320(8):825-833. doi: 10.1001/jama.2018.10574. PMID 30167704